CLINICAL TRIAL: NCT06082544
Title: Clinical And Radiographic Success Of Mini Screw Implant Supported Pontics Versus Removable Partial Dentures For Restoring Missing Permanent Anterior Teeth: Randomized Clinical Trial
Brief Title: Mini Screw Implant Supported Pontics Versus Removable Partial Dentures For Restoring Missing Permanent Anterior Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Adel Abd Elhameed, assistant lecturer in the department of pediatric dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 29208130101509
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Missing Teeth
MeSH Terms: conditions — Anodontia | interventions — Denture, Partial, Removable

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mini-screw implant-supported pontics placed palatally perpendicular to the alveolar ridge (Experimental): Mini-screw implant-supported pontics placed palatally perpendicular to the alveolar ridge (horizontally placed) using JEIL SCREW 1.6*8 MM 16-G2-008
  Interventions: Other: mini-screw implant
- Mini screw implant supported pontics placed at the crest of the ridge (Experimental): Mini screw implant supported pontics placed at the crest of the ridge (vertically placed) using JEIL SCREW 1.6* 10 MM 14-G2-f010
  Interventions: Other: mini-screw implant
- Removable partial denture. (Active Comparator): removable partial denture with conventional technique
  Interventions: Device: removable partial denture

INTERVENTIONS:
Other: mini-screw implant — JEIL SCREW 1.6* 8 MM 16-G2-008 or JEIL SCREW 1.6*10 MM 14-G2-010
  Arms: Mini screw implant supported pontics placed at the crest of the ridge; Mini-screw implant-supported pontics placed palatally perpendicular to the alveolar ridge
Device: removable partial denture — Acrylic removable partial denture
  Arms: Removable partial denture.

SUMMARY:
Loss of teeth leads to loss of function and lack of normal alveolar growth, along with unpleasant esthetics that hamper the psychosocial development of the young child. Traditionally, the management of single tooth loss in a young child is done by conservative means. The presence of large pulp chambers in incompletely mineralized immature teeth of children predisposes the pulp to loss of vitality in cases of complete coverage restorations . Hence, the clinician resorts to partial coverage prostheses such as Maryland Bridge, resin-bonded restorations, or removable prostheses in cases of multiple missing teeth. None of these treatment methods are completely satisfactory and have their drawbacks.

Partial dentures are dependent on the child's compliance. They increase the rate of decay and may cause gingival disease leading to bone resorption. Furthermore, there is a need to refabricate a new prosthesis from time to time to compensate for craniofacial growth.

Mini-screw implant placement in a young child would be an ideal method of treatment for the absence of teeth. They restore the function, preserve the alveolar bone, and give excellent esthetics, restoring the child's confidence and social acceptability. Parents are usually keen to get this treatment done as soon as offer the suggestion. To our knowledge, there is no previous study that compared the two techniques. The limited evidence shows that mini-screw implants supported pontics are useful transitional restorations for missing permanent maxillary incisors in children and adolescents; however, further well-designed clinical trials are needed in this regard. As a result, this study will be conducted to fill the gap of knowledge.

DETAILED DESCRIPTION:
Rationale for conducting the research Mini- screw implant prosthetic rehabilitation seems to be a viable and promising option for provisional rehabilitation of growing patients, since it seems to preserve the bone structure while restoring function and esthetics until growth ceases, when then mini-screw implants can be replaced by standard implants.

Benefits for the practitioner:

* Providing new and alternative treatment options for restoring missing permanent anterior teeth with fixed mini-screw implant supported pontics.
* Increasing the compliance of the patients.

Benefits for the patient:

* Re-establish esthetic and appearance.
* Maintenance of space.
* Re-establishing occlusal relationships.
* Improving phonetics.
* Improving patients tolerance.
* Improvement in patient as well as parent satisfaction.

Benefits for community:

* Using alternative technique that can be fixed, with a better success rate.
* To boost overall oral health.

ELIGIBILITY:
Inclusion Criteria:

* • Cooperative children.

  * 9:14 years old children.
  * Children with missing anterior permanent teeth either due to caries, trauma (at least 4 months after missing the tooth) or congenitally missed.

Exclusion Criteria:

* Children with physical or emotional alteration.
* Children with systemic diseases.
* Children of parents who don't accept to participate in the study.
* Very thin ridge

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 3,6,9,12 months
  visual analogue scale (VAS) continuous from 0-10 (0 not satisfied at all and 10 is satisfied)
adverse effects | 3,6,9,12 months
  denture fracture, denture loss, denture remake, looseness of the screw, fracture of the screw, pontic displacement, fracture of the pontic and discoloration of the pontic

SECONDARY OUTCOMES:
vertical bone resorption | 1 year
  parallel technique using periapical radiograph
horizontal bone resorption | 1 year
  Cone beam computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Eman A Abdelhameed, MD, Principal Investigator — Assistant lecturer at Pediatric Dentistry and Dental Public Health Department; Gihan M Abuelniel, PHD, Study Director — Professor at Pediatric Dentistry and Dental Public Health Department; Ahmed H El Khadem, PHD, Study Director — Associate Professor at Pediatric Dentistry and Dental Public Health Department; Maii M Mohamed, PHD, Study Director — Lecturer at Pediatric Dentistry and Dental Public Health Department; Ahmed M Abdel Samad, PHD, Study Director — Professor at Oral and Maxillofacial Radiology Department
Locations (1):
- Faculty of Dentistry, Cairo University, Giza, Al Manial, Egypt